CLINICAL TRIAL: NCT06425887
Title: Smartwatch Paroxysmal Arrhythmia Detection Compared with Holter - a Multicenter Controlled Trial
Brief Title: Smartwatch Paroxysmal Arrhythmia Detection Compared with Holter
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: Smartwatch vs Holter study
Record Dates: First submitted 2024-05-03; First posted 2024-05-23 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-05

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Smart watch — not interventional

SUMMARY:
The lifetime risk for development of atrial fibrillation, the commonest sustained arrhythmia in adults, is estimated to be 24%-27% for individuals of 40 years or older. Previous work showed that annual new diagnosis of AF is 11000-26000 in Hong Kong. Other arrhythmia such as supraventricular arrhythmia or premature beats were also common and of clinical significance.

12-lead ECG is a first line investigation for patients with suspected paroxysmal arrhythmia, but it has a low diagnostic yield with its 10-30 seconds recordings. 24-hour Holter exam is the usual next step of diagnosis. The diagnostic yield of Holter varies according to indication but is generally low at 1%-12%. This is because paroxysmal arrhythmia may not happen every day. In addition, even if arrhythmia is picked up in Holter, patient may not register the symptom, making the symptom arrhythmia correlation problematic.

Despite limitations, the demand for Holter exam is still high. In Prince of Wales Hospital, a tertiary referral centre with a catchment of about 1 million populations, the waiting time for a routine Holter exam is 3 years.

Smartwatch has gained popularity over past years as an adjunct to smartphone. Latest generations of smartwatch were equipped with wearer-initiated ECG rhythm strip recording capabilities. Smartwatch has evolved to become a health tracker with arrhythmia detection capabilities. It was found to be a useful tool for atrial fibrillation screening in general population. Other arrhythmias, such as supraventricular tachycardia, premature beats, and abnormal ECG patterns associated with sudden cardiac death could also be detected with smartwatch ECG recordings. Apple Heart study was the largest study utilizing smartwatch for arrhythmia detection. The general population was screened for atrial fibrillation using irregular pulse algorithm. The study found a 84% concordance rate between irregular pulse notification and ECG patches.

Therefore, investigators propose to conduct a study to compare its diagnostic yield with Holter, in patients with suspected arrhythmia and see if smartwatch recording following a systematic protocol for four-weeks will have better arrhythmia diagnosis yield than a 24-hour Holter exam.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred for out-patient Holter exam from age 18 - 80 years old
2. The following indications for Holter exam will be allowed for recruitment

   * Palpitation
   * Pre-syncope
   * Dizziness

Exclusion Criteria:

1. Patients with a prior ECG diagnosis to explain the symptom
2. Primary symptom is syncope
3. Patient who has no clear indication for Holter exam
4. Pregnant ladies
5. Patients who failed to make a successful recording despite teaching attempts.
6. Patients who cannot read English or Chinese version of consent.
7. Anticipation of non-compliance with recording protocol.
8. Patients who do not have a compatible smart phone (Android 9.0 or newer, or iOS15 or newer)
9. Patients under custody

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being referred for out-patient Holter exam will be reviewed for eligibility. Individuals aged 18 to 80 with indications for Holter including palpitation, pre-syncope & dizziness without meeting any exclusions will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison | through study completion, an average of 1 month
  Compare the percentage of patients with significant arrhythmia diagnosed, between smartwatch rhythm recording and 24-hour Holter arm Significant arrhythmia is defined as the presence of any one of the following
  * Sustained supraventricular tachycardia (>=30 seconds)
  * Atrial fibrillation (>=30 seconds)
  * Ventricular tachycardia of more than 3 consecutive beats
  * Significant AV block (defined as 2nd degree Mobitz type II or 3rd degree heart block)
  * HR less than 40 while awake.
  * Pause > 2 seconds while awake (for both smartwatch and Holter), or >3 seconds while asleep (for Holter only)
  * Premature ventricular complex with an overall burden of more than 10%

SECONDARY OUTCOMES:
Detection rate | through study completion, an average of 1 month
  describe the detection rate of smartwatch for various arrhythmia
Preference | through study completion, an average of 1 month
  describe patients' preference on using which modality (smartwatch or Holter) to record their arrhythmia, by means of a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No